CLINICAL TRIAL: NCT04260100
Title: The Effects of Diabetic Care Self-Management Mobile Health Application on Foot Care Behaviour, Dietary Behaviour, Foot Conditions and Fasting Blood Glucose Among Diabetes Mellitus Clients in Malaysia
Brief Title: Diabetic Care Self-Management Mobile Health Application Among Diabetes Mellitus Clients in Malaysia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohd Khairul Zul Hasymi Firdaus (Other)
Collaborators: Prince of Songkla University (Other)
Responsible Party: Sponsor-Investigator, Mohd Khairul Zul Hasymi Firdaus, Sponsor-Investigator, Prince of Songkla University
Organization: Prince of Songkla University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Diabetic Care Mobile App
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Diabetes Care Self-Management Mobile Health Application
- Control Group (No Intervention): Routine care group

INTERVENTIONS:
Behavioral: Diabetes Care Self-Management Mobile Health Application — In day 1, the participant will receive a Foot Care Kit consist of a mirror, a tube of lotion, a small towel, and a nail clipper. The participant will enrol in 3-hour workshop for general management of diabetes mellitus, diabetic foot care and dietary management. The participant will be invited to install Diabetes Care Self-Management Mobile Health Application. The mobile application is meant for sources of referral for diabetic foot care and dietary care, and for record purpose (diary) of any foot care activities carried out that participant needs to enter in the application during his/her home. The participant will be trained for the use of Diabetes Care Mobile Health Application. In addition, the participant will be invited to join a WhatsApp group for the medium of communication. The program will be lasting for 5 weeks.
  Arms: Intervention Group

SUMMARY:
The main purpose of this study is to explore the effect of Diabetic Care Self-Management Mobile Health Application in behavioral modification i.e foot care behaviour and dietary behaviour among diabetic clients in Malaysia. Diabetic Care Self-Management Mobile Health Application is a mobile health (mHealth) application program aiming for primary care in health prevention and promotion activity. The program is developed by the researcher through the literature review conducted. The program is evaluated through a randomized controlled trial study design.

ELIGIBILITY:
Inclusion Criteria:

* Past readings of A1c more than 6.5% (Ministry of Health Malaysia, 2015).
* Has at least Stage 1 or above for the risk of foot ulcer development. The risk will be identified through diabetic foot screening. The screening will be carried out by using Inlow's 60 Second Diabetic Foot Screen.
* Age of 18 to 65 years old. Since the study is using mobile health applications, technology literate is an important factor to see the effect of mHealth on behaviour modification process. If the patient is more than 65 years old, the patient might have some difficulties in using mobile health intervention. Meanwhile, for the patient less than 18 years old, guardian permission is required prior to study enrolment.
* Have no history of diabetic foot ulcers.
* Able to independently perform self-care.
* Able to use a mobile application program.
* Own an android phone.
* No vision or hearing problem may interfere with the process of data collection and intervention carried out.
* Able to communicate in either English or Bahasa Malaysia (a native and official language of the country)

Exclusion Criteria:

* The patient that did not come for the follow-up care at Week 5. For instance, the patient may have other matters on the day of follow-up up which required their urgent attention and not able to come for the follow-up, or is stay outside of the area during the day of follow up.
* Have difficulty in performing foot care during in the middle of the intervention period. For example, the client may get sick due to hypoglycemic or hyperglycemic attack which stopped them from being able to perform the foot care behaviour.
* The patient is diagnosed with any cognitive and perceptual decline function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Foot Care Behaviour | 5 weeks; Baseline on Week 1 and follow up on Week 5
  The changes of foot care behaviour will be measured twice (Week 1 and Week 5) by using Diabetic Foot Selfcare Behaviour Scale (DFSBS). The questionnaire consist of two parts namely Part 1 and Part 2 with two set of different responses. In Part 1, there are four different questions measuring the self-care activity. The response for this Part 1 consists of days performed from 0 - 7 days. The response will be categorized based on Likert Scale according to the following categories; 0 days for score of 1, 1-2 days for score of 2, 3-4 days for score of 3, 5-6 days for score of 4 and 7 days for score of 5. In Part 2, the question responses are categorized as never (1), seldom (2), sometimes (3), frequently (4) and always (5). The total score accumulated will be in range of 7 - 35. The interpretation of the score will be the higher the score, the better the foot care behaviour.
Dietary Behaviour | 5 weeks; Baseline in Week 1 and follow up in Week 5
  The changes of dietary behaviour will be measured twice (Week 1 and Week 5) by using translated Dietary Behavior Questionnaire (DBQ). The questionnaire consists of 30 items with four domains. The domains are selecting a healthy diet with 13 items; arranging a meal plan, 7 items; recognizing the amount of calorie needs, 5 items and managing dietary behaviour challenges, 5 items. 5 points of Likert scale is use from 0 to 4 with 0 for never, 1 for seldom, 2 for occasionally, 3 for often and 4 for repeatedly. The total score of DBQ is ranging from 0 to 120 with score of 0 to 40 categorized as poor behaviour, 41 to 80 categorized as medium and 81 to 120 categorized as better dietary behaviour.

SECONDARY OUTCOMES:
Foot Conditions | 5 weeks; baseline in Week 1 and post intervention in Week 5
  The foot conditions will be assessed twice (Week 1 and Week 5) by using foot condition assessment form.
Fasting Blood Glucose | 5 weeks; baseline in Week 1 and post intervention in Week 5
  The level of fasting blood glucose will be assessed twice (Week 1 and Week 5) by withdrawing participants blood for the test.The test will be sent to a certified laboratory for the analysis of FBG reading. Prior to blood taking procedure, the participants will be asked to fast.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Kesihatan UTC Kangar, Kangar, Perlis Indera Kayangan, Malaysia

REFERENCES:
- [Derived] Firdaus MKZH, Jittanoon P, Boonyasopun U, Che Hasan MK. The effect of mHealth program on behavior modification and health outcomes among patients with diabetes: A randomized controlled trial study. Belitung Nurs J. 2023 Oct 26;9(5):437-447. doi: 10.33546/bnj.2664. eCollection 2023. PMID 37901368